CLINICAL TRIAL: NCT02216669
Title: Phase I Trial to Determine Optimal Phase II Dose of the Oral Dual CAIX Inhibitor/ Radiosensitizer
Brief Title: Trial to Determine Optimal Phase II Dose of the Oral Dual CAIX Inhibitor/ Radiosensitizer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No financial agreement
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-2014
Record Dates: First submitted 2014-08-08; First posted 2014-08-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Solid Tumors; Head and Neck Neoplasms
Keywords: Solid tumors; Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DTP348 (Experimental): Patients will receive a continuous oral dose of DTP348 for 7 days per week for 7 weeks
  Interventions: Drug: DTP348

INTERVENTIONS:
Drug: DTP348 — Patients will receive a continuous oral dose of DTP348 for 7 days per week for 7 weeks
  Other Names: 2-(2-methyl-5-nitro-1H-imidazol-1-yl)ethylsulfamide

SUMMARY:
This is a Phase I multicenter, open-label, dose-escalation study of DTP348. DTP 348 is an oral dual drug with two mechanisms of action:

1. carbonic anhydrase IX inhibitor which acidifies the intracellular pH through the sulfamide components
2. radio sensitizer of hypoxic cells through its 5-nitroimidazole moiety

The study will be conducted in 2 parts. The phase I trials will be on the standard 3+3 design first as single agent then combined with radiotherapy:

1. A single agent dose-escalation phase in patients with solid tumours.
2. A dose-escalation phase in patients with HNSCC in combination with radiotherapy

The main objective is to determine the recommended phase II dose of DTP348 in combination with radiotherapy

DETAILED DESCRIPTION:
In the single agent Phase I dose-escalation phase patients will be enrolled and assigned to a dose level cohort. The starting dose will be 750 mg/m2, which equals to 1/10 of the human equivalent dose of the LD10 of DTP348 in mice.

A "3+3" dose-escalation design will be used. The study will investigate sequential cohorts consisting of 3-6 patients to be enrolled and treated at the applicable dose level. Planned dose levels for subsequent cohorts are 1000, 1250 mg/m2 and steps of 250 mg/m2 thereafter. There will be no intra-patient dose escalation. The treatment cycle in the dose-escalation part of the study will consist of 7 weeks (reflecting the typical duration of the course of radiotherapy). Patients will receive a continuous oral dose of DTP348 for 7 days per week. Food intake is not allowed one hour before and after the intake of the study drug. After the cycle of treatment, the patient will be followed until disease progression.

Blood samples for pharmacokinetic properties (PK) will be obtained on day 1 during the first 8 hours after oral administration and then daily on day 2, 3, 4 and 5, before the administration of the daily dosage. A patient will stay on treatment until disease progression, unacceptable toxicity, or discontinuation for any other reason. The dose limiting toxicity (DLT) observation period for each dose level will be day 1 until the end of week 7. Patients who do not complete the DLT observation period for other reasons than a DLT will be replaced.

Toxicity that can be expected from DTP348 is related to the nitro-imidazole compound and includes nausea, vomiting flushing, dizziness, skin rash, and neurotoxicity. Related to the sulfamide component in the study drug, the side-effects may include nausea and vomiting. In the experimental mice study, no toxicity was observed using a dose of 10 mg/kg i.v. 3 and up to 400 mg/kg per os, which corresponds to the Human Equivalent Dose (HED) of 1.2 g/m2 of nimorazole. Once the Maximum Tolerated Dose (MTD) of DTP348 has been established, 3 additional patients will be included in that dose-level. These patients will receive crushed tablets and undergo blood sampling for PK to investigate whether the administration of crushed tablets affects uptake and plasma levels of the study drug. This group of patients is added because of the frequent occurrence of swallowing problems in the HNSCC patient population and the use of tube feeding with the need of crushing tablets.

Once the MTD of DTP348 as single agent has been determined, the study will continue to the combination phase: In the DTP348 in combination with radiotherapy dose-escalation phase, again a 3+3 dose-escalation design will be used. The starting dose of DT348 will be the MTD minus two dose levels. DTP348 will be given continuously 7 days a week, starting 2 weeks before and during the whole course of radiation until and including the last day. The rationale to start the study drug 2 weeks before the start of radiotherapy is to have a similar design as in the phase II trial which will be performed following this study. The drug will be given orally 1-2 hours before the daily delivery of radiotherapy. Food intake is not allowed one hour before and after the intake of the study drug. The dose limiting toxicity (DLT) observation period for each dose level will be from day 1 of combined therapy until 4 weeks after the end of therapy. Patients who do not complete the DLT observation period for other reasons than a DLT will be replaced.

The radiation treatment in the DTP348 in combination with radiotherapy dose-escalation phase will be either conventional standard fractionated radiotherapy to a total dose of 70 Gy in 35 fractions over 7 weeks with a concomitant boost technique, 5 fractions a week or accelerated radiotherapy delivering a total dose to 68-70 Gy in a shortened overall treatment time (5.5 - 6 weeks). The 95% isodose of the prescribed dose should encompass at least 99% of the planning target and homogeneity will be according to ICRU guidelines. There is no restriction of the treatment techniques that may be used: multiple static conformal or intensity modulated beams, intensity modulated arc treatments, or robotic, non-isocentric treatments. Dummy run on virtual patients will need to be performed before inclusion. Subsequently, patients are allowed to be included in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative measures or other therapy that may provide clinical benefit do not exist or are no longer effective.
* Age 18 year or older
* Performance status, WHO = 0 - 2
* Subject must have adequate bone marrow, renal and hepatic function per local laboratory reference rage as follows:

Bone marrow: absolute neutrophil count (ANC) >/= 1,500/ul; platelets >/= 100,000/mm3 (independent of platelet transfusion, within 3 months prior to starting study drug); haemoglobin >/= 9.0 g/dL

Renal function: serum creatinine </= 2.0 mg/dL or calculated creatinine clearance >/= 50 mL/min

Hepatic function and enzymes: AST and ALT </= 2.5 x the upper limit of normal (ULN) of institution's normal range. Bilirubin </=1.5 x INL.

Subjects with liver metastases may have an AST and ALT of </= 5.0 x ULN

* Measurable disease (RECIST, version 1.1)
* Subjects with known brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and or radiation therapy followed by 21 days of stable neurologic function and no evidence of CNS disease progression as determined by comparing a computed tomography (CT) scan or magnetic resonance imaging (MRI) scan performed during screening to a prior scan performed at least 4 weeks earlier and provided that the subject is asymptomatic, has no evidence of cavitation or haemorrhage and is on a stable dose of dexamethasone.
* Females must have negative results for pregnancy tests performed:

At screening on a serum sample obtained within 7 days prior to initial study drug administration, and Prior to dosing on a urine pregnancy test will be obtained prior to study drug administration (cycle 1, day 1).

* No breast feeding.
* If female, subject must be either postmenopausal for at least 2 years, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or practicing at least one of the following methods of birth control:

Total abstinence from sexual intercourse as the preferred life style of the subject, periodic abstinence is not acceptable; Vasectomized partner; Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration (if the subject is currently using a hormonal contraceptive, she should also use a barrier method during the study and for 1 months after study completion); Intrauterine device (IUD); Double barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or creams);

- If male, subject must be surgically sterile or practicing at least 1 of the following methods of contraception and refrain from sperm donation, from initial drug administration until 90 days after the last dose of study drug: Partner(s) using an IUD; Partner(s) using hormonal contraceptives (oral, vaginal, parenteral or transdermal); Subject and/or partner(s) using double-barrier method (condoms, contraceptive sponge, diaphragm, or vaginal ring with spermicidal jellies or creams).

Total abstinence from sexual intercourse as the preferred life style of the subject; periodic abstinence is not acceptable.

* Ability to swallow and take oral medication. Patients that are dependent on a feeding tube can only be included in the study when entered in the last cohort, in which the PK of crushed study medication is the object of study.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Willing and able to undergo blood sampling for pharmacokinetics
* Must voluntarily sign and date each informed consent, approved by an independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* If the subject has clinically significant and uncontrolled major medical condition(s) including but not limited to:

Uncontrolled seizure disorder, including focal or generalised seizure within the last 12 months; Uncontrolled nausea/vomiting/diarrhea; Active uncontrolled infection, including HIV and hepatitis (HBV, HCV) Symptomatic congestive heart failure, irreversible cardiac arrhythmias, acute or subacute coronary syndromes within the last year.

Psychiatric illness/social situation that would limit compliance with study requirements Any medical condition, with the opinion of the study investigator, places the subject at an unacceptably high risk for toxicities.

* Female subject is pregnant or breastfeeding.
* Subject has received any of the following anti-cancer therapies 21 days prior to the first dose of study drug:

Chemotherapy, immunotherapy, radiotherapy.

Any investigational therapy, including targeted small molecule agents. With the following exceptions:

* Hormonal anticancer therapy must be stopped 7 days before starting day 1 of cycle 1 (C1D1)
* Hormones for hypothyroidism, estrogen replacement therapy (ERT) or agonists required or suppress serum testosterone or estrogen levels (e.g. LHRH, GnRH, etc) for subjects with prostate, breast and ovarian cancer if on a stable dose for 21 days prior to the first dose of study drug.
* Subject has received a biological agent for anti-neoplastic intent within 30 days prior to the first dose of study drug.
* Subject who requires parenteral nutrition, tube feeding or has evidence of partial bowel obstruction or perforation within 28 days prior to study drug administration.
* The subject has had another active malignancy within the past 3 years except for any cancer in situ that the Principal Investigator considers to be cured.
* In the opinion of the investigator, the subject is an unsuitable candidate to receive DTP348.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The maximum-tolerated dose (MTD) of DTP348 as single agent | 3 months
  To assess the safety and tolerability of DTP348 when administered orally as single agent in patients with advanced solid tumours in order to determine the Maximum Tolerated Dose (MTD) in relation with the occurrence of a Dose Limiting Toxicity (DLT).
The maximum-tolerated dose (MTD) regimen of DTP348 as single agent in combination with radiotherapy | 3 months
  To assess the safety and tolerability of DTP348 when administered orally in combination with radiotherapy in patients with HNSCC and to determine the Recommended Phase II Dose (RP2D) of this treatment combination.

SECONDARY OUTCOMES:
Plasma concentration of DTP348 | 3 months
  To characterise the Pharmacokinetic (PK) properties of DTP348 after oral administration as single agent
Response rate according to RECIST, version 1.1, DTP348 monotherapy | 3 months
  To evaluate the preliminary efficacy of DTP348 monotherapy in terms of anti-tumour activity
Response rate according to RECIST version 1.1, DTP348 in combination of radiotherapy | 3 months
  To evaluate the preliminary efficacy of DTP348 in combination with radiotherapy in terms of anti-tumour activity in patients with HNSCC.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hoebers, Dr., Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastro Clinic, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No